CLINICAL TRIAL: NCT07283081
Title: Impact of Capillaroscopy in the Investigation of Diffuse Interstitial Pneumonias
Acronym: CAPID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2025/086
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Interstitial Lung Disease; Connective Tissue Diseases
Keywords: Pulmonary Interstitial Disease; capillaroscopy; Connective Tissue Disease; diagnosis
MeSH Terms: conditions — Lung Diseases, Interstitial; Connective Tissue Diseases; Disease | interventions — Microscopic Angioscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diffuse interstitial lung diseases (DILD) (Experimental)
  Interventions: Diagnostic Test: capillaroscopy

INTERVENTIONS:
Diagnostic Test: capillaroscopy — Capillaroscopy will be performed during a specific consultation. During this examination, a device called a "video capillaroscope" is used to magnify and visualize the capillaries located at the base of the nail. The examination lasts approximately twenty minutes.

SUMMARY:
The investigators hypothesize that in patients with a new diagnosis of Pulmonary Interstitial Disease (PID), adding capillaroscopy to standard care increases the proportion of patients receiving a diagnosis of PID-Connective Tissue Disease (PID-CTD) within the first three months of follow-up, thereby reducing the time to diagnosis and facilitating the implementation of appropriate treatment as quickly as possible. Therefore, To confirm this hypothesis, it is necessary to know the characteristics of capillaroscopy in patients with a new diagnosis of PID.

DETAILED DESCRIPTION:
Diffuse interstitial lung diseases (DILD) are a group of diseases characterized by inflammation and fibrosis of the lung tissue, with more than 200 identified causes, approximately 20% of which are related to autoimmune diseases such as connective tissue disorders (e.g., scleroderma, lupus). Pulmonary involvement may precede the diagnosis of connective tissue disease, making diagnosis difficult. Capillaroscopy, a non-invasive and reproducible test, is used to detect microvascular abnormalities, especially in scleroderma spectrum diseases, but its precise role in the evaluation of PID is still poorly defined. Studies show that PIDs associated with autoimmunity are more likely to present with capillaroscopic abnormalities. However, current recommendations on the investigation of PIDs do not clearly specify the use of capillaroscopy, and there are no studies establishing its value in systematic screening of all patients with PID. Thus the investigators aim to describe the characteristics of capillaroscopy in patients with a new diagnosis of PID.

The project will be offered to eligible patients for whom a PID has been identified. A review of the medical record information will then be carried out, with additional tests performed as necessary to identify the etiology associated with this IDP. The compilation of information, and especially the performance of additional tests (beyond normal care), is typically completed within three months. In the meantime, and particularly in the first month after signing the consent form, the patient will undergo a capillaroscopy and complete the patient questionnaire. After three months, once all additional tests have been performed and the results compiled, the pulmonologist completes the questionnaire to identify the most likely etiology of the patient's PID. All tests, except for capillaroscopy, are performed as part of routine care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years of age;
* Have received a new diagnosis of PID within the last six months, confirmed by a pulmonologist;
* Have undergone some specific tests within the last six months (Chest CT scan, respiratory function tests (plethysmography and CO transfer capacity measurement, immunological assessment including: screening for FAN, FR, and anti-CCP);
* French-speaking patient with no comprehension difficulties;
* Person affiliated with or beneficiary of a social security system;
* Free, informed, and written consent signed by the participant and the investigator (no later than the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Have previously undergone a capillaroscopy, regardless of the reason;
* Have a diagnosis or high suspicion of connective tissue disease based on initial clinical and paraclinical evaluation;
* Have already started one of the following treatments for pulmonary involvement: systemic corticosteroids, immunosuppressive therapy, antifibrotic therapy;
* Pregnant or breastfeeding women;
* Patients covered by Articles L 1121-5 to L 1121-8 (persons deprived of their liberty by judicial or administrative decision, minors, adults subject to legal protection measures, or persons unable to give their consent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of capillaroscopy abnormalities according to the classification proposed by the EULAR Study Group on Microcirculation in Rheumatic Diseases | At baseline (Day 0)

SECONDARY OUTCOMES:
Description of the criteria that may influence the results of capillary examination: proportion of smoking status categories (active smoker/non-smoker/former smoker) and number of cigarettes per day for active smokers | At baseline (Day 0)
Description of the criteria that may influence the results of capillary examination: number of cigarettes per day for active smokers | At baseline (Day 0)
Description of the criteria that may influence the results of capillary examination: proportion of patients who consume alcohol | At baseline (Day 0)
Description of the criteria that may influence the results of capillary examination: average number of standard drinks for active consumers. | At baseline (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Elise TRUCHETET, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - service de rhumatologie, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No